CLINICAL TRIAL: NCT03583931
Title: Early Intervention for Complicated Parapneumonic Effusion: Randomized Controlled Trial for Fibrinolytic Therapy Versus VATs Decortication
Brief Title: Treatment of Complicated Parapneumonic Effusion With Fibrinolytic Therapy Versus VATs Decortication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0857
Record Dates: First submitted 2018-05-11; First posted 2018-07-12 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2021-11

CONDITIONS: Parapneumonic Effusion; Empyema, Pleural; Coagulopathy
Keywords: VATS Decortication; Surgical Pleural Decortication; Fibrinolytic Therapy; Pneumonia; Thoracostomy
MeSH Terms: conditions — Empyema, Pleural; Hemostatic Disorders; Pneumonia | interventions — Thrombolytic Therapy; Deoxyribonucleases

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Clinical Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operative VATS decortication (Active Comparator): Operative group that will undergo early VATS decortication of complicated parapneumonic effusion/empyema
  Interventions: Procedure: VATS Decortication
- Non-operative Fibrinolytic Therapy (Active Comparator): Non-operative group that will undergo instillation of the drugs DNAse and tPA (tissue plasminogen activator) together i.e. 5mg DNAse and 10mg tPA twice a day for up to six doses, through chest tube as treatment of the patient's complicated parapneumonic effusion/empyema. Fibrinolytic therapy = DNAse + tPA; these medications are not mutually exclusive.
  Interventions: Drug: Fibrinolytic Therapy

INTERVENTIONS:
Procedure: VATS Decortication — Surgical procedure to unroof all located collections of the pleural space through a chest wall incision
  Arms: Operative VATS decortication
Drug: Fibrinolytic Therapy — Instillation of DNAse and tPA together through patient's chest tube already in placed to break down complex fluid collection in the pleural space. DNAse and tPA are are administered together only i.e. are not mutually exclusive.
  Other Names: DNAse / tPA combination therapy.
  Arms: Non-operative Fibrinolytic Therapy

SUMMARY:
This study aims to standardize the treatment of pleural space (parapneumonic) infections by comparing the difference in outcomes between 2 methods of treatment: early VATS (Video Assisted Thorascopic Surgery) decortication versus fibrinolytic therapy. During treatment, the patient's coagulopathy status will also be evaluated.

DETAILED DESCRIPTION:
The treatment of parapneumonic infections (infection in the pleural space) at the Denver Health Medical Center is not standardized, and timing for advanced interventions such as fibrinolytic therapy or surgical decortication remain unclear. The definitive treatment strategy in these patients may be sub-optimal, and lead to prolonged hospitalization and morbidity. This is concerning as the mortality rate of community acquired pneumonia triples in the presence of a parapneumonic process (5-15%) and can reach over 25% if it becomes bilateral(1). Prompt recognition of pleural space infections is essential for reducing morbidity and mortality. This is attributable to the progression of the disease from a simple fluid collection amenable to pleural space drainage, to necrotizing empyema requiring thoracotomy decortication and open drainage. The keys to management of parapneumonic effusions are early diagnosis, appropriate therapeutic intervention, and recognition of failure of conservative management. The investigators propose that a standardized pathway for identifying and treating parapneumonic effusions will be an important quality improvement. A key gap in the literature remains if patients with parapneumonic infections that cannot be drained with a chest tube should undergo a trial in intrapleural fibrinolytic therapy, or if they should go directly to video assisted thoracic surgery (VATS) for decortication of all infectious material.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Admitted with pleural effusion that undergoes thoracentesis by medical/pulmonary service
* Pleural fluid pH <7.3
* SICU placed chest tube
* Subsequent transfer to SICU

Exclusion Criteria:

* Existing malignancy
* Malignant cells from initial pleural fluid sample
* End stage liver disease (Child's B or greater)
* Coagulopathy
* Unable to tolerate surgical procedure
* Frank purulent drainage (needs OR regardless)
* Recent surgery of abdomen or thorax precluding the use of tPA
* Baseline neurologic impairment requiring a proxy for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredric Pieracci, MD, MPH, Principal Investigator — Denver Health and Hospital
Locations (1):
- Denver Health, Denver, Colorado, United States

REFERENCES:
- [Derived] Barrett CD, Moore PK, Moore EE, Moore HB, Chandler JG, Siddiqui H, Maginot ER, Sauaia A, Perez-Calatayud AA, Buesing K, Wang J, Davila-Chapa C, Hershberger D, Douglas I, Pieracci FM, Yaffe MB. Neutrophil-Mediated Inflammatory Plasminogen Degradation, Rather Than High Plasminogen-Activator Inhibitor-1, May Underly Failures and Inefficiencies of Intrapleural Fibrinolysis. Chest. 2025 Jan;167(1):67-75. doi: 10.1016/j.chest.2024.04.005. Epub 2024 May 6. PMID 38710463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective randomized clinical trial of hospitalized patients identified to have complicated parapneumonic effusions with radiographic imaging. Denver Health and Hospital Authority.
Period: Overall Study
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 subjects were enrolled. Five were randomized to the FT group and 5 to early VATS decortication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (16.1) | 45.6 (11.1) | 44.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: How long the patient remains admitted in the hospital during their index hospitalization
Time Frame: From patient's admission to hospital to their discharge, (excluding extended stay due to social work reasons) up to 28 days or discharge, which ever comes first.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
days | 12.4 (16.7) | 8.4 (4.1)

2. Secondary Outcome: ICU Free Days
Description: Admission days during index hospitalization that are of a lower acuity of care than intensive care
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: All 10 participants were analyzed on this data point and aggregate data is provided below for each treatment arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
Days | 22.4 (8) | 20 (6.2)
Statistical Analysis 1: Comparison: Operative VATS Decortication vs Non-operative Fibrinolytic Therapy; Test type: Superiority; p = 0.61, ANOVA

3. Secondary Outcome: Chest Tube Days
Description: Days with chest tube in place after intervention
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: All 10 participants were analyzed on this data point and aggregate data is provided below for each treatment arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
Days | 7.4 (8.2) | 8.2 (2.4)
Statistical Analysis 1: Comparison: Operative VATS Decortication vs Non-operative Fibrinolytic Therapy; Test type: Superiority; p = 0.84, ANOVA

4. Secondary Outcome: Cost of Admission and Treatment
Description: Cost of care for the patient after their intervention
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: The data were not collected
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pain Score
Description: What the patient's level of pain is from 0 to 10; zero being no pain, 10 being the worst pain imaginable. score is categorical 0,1,2,3,4,5,6,7,8,9 or 10.
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: The pain score was provided at the discharge date or at 28 days of admission (whichever came first).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 4 | 5
score on a scale | 3.6 (1) | 4.6 (2)

6. Secondary Outcome: Chest Tube Drainage
Description: The amount and character of the drainage from the chest tube after intervention
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: Incomplete analysis documented in records on this measure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 4 | 5
mL | 60.1 (12.3) | 713.2 (180.3)

7. Secondary Outcome: Incentive Spirometry
Description: To what volume the patient can inspire using an incentive spirometer
Time Frame: Everyday for 5 days post study intervention, from admission to discharge, or for 28 days, whichever comes first.
Population: No participants were analyzed on this measure in the final analysis, because the data were not collected.
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Supplemental Oxygen Days
Description: The amount of time the patient needs to warn off any supplemental oxygen
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: All 10 participants were analyzed on this data point and aggregate data is provided below for each treatment arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
Days | 17.8 (24.5) | 9.6 (2.3)
Statistical Analysis 1: Comparison: Operative VATS Decortication vs Non-operative Fibrinolytic Therapy; Test type: Superiority; p = 0.48, ANOVA

9. Secondary Outcome: Fever Days
Description: The amount of days it takes to resolve fever (temp >100.4)
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: All 10 participants were analyzed on this data point and aggregate data is provided below for each treatment arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
Days | 4.8 (5.3) | 0.8 (1.1)
Statistical Analysis 1: Comparison: Operative VATS Decortication vs Non-operative Fibrinolytic Therapy; Test type: Superiority; p = 0.25, ANOVA

10. Secondary Outcome: Days of Antibiotics
Description: The number of days antibiotics are required after intervention
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: All 10 participants were analyzed on this data point and aggregate data is provided below for each treatment arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
Days | 17 (9.3) | 25.6 (24.6)
Statistical Analysis 1: Comparison: Operative VATS Decortication vs Non-operative Fibrinolytic Therapy; Test type: Superiority; p = 0.45, ANOVA

11. Secondary Outcome: Elevated White Blood Count Days
Description: The amount of days it takes to resolve a leukocytosis
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: All 10 participants were analyzed on this data point and aggregate data is provided below for each treatment arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 5 | 5
Days | 5.6 (4) | 6 (3.6)
Statistical Analysis 1: Comparison: Operative VATS Decortication vs Non-operative Fibrinolytic Therapy; Test type: Superiority; p = 0.87, ANOVA

12. Secondary Outcome: Changed in Coagulopathic Status
Description: Changes in laboratory TEG values after intervention
Time Frame: From admission to discharge, or for 28 days, whichever comes first.
Population: No participants were analyzed on this measure in the final analysis, because the data were not collected.
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, average of 1 year, which was the length of time participants were followed.
Arm/Group | Operative VATS Decortication | Non-operative Fibrinolytic Therapy
All-Cause Mortality (participants affected / at risk) | 0/5 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/5
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Operative VATS Decortication (N=5) | Non-operative Fibrinolytic Therapy (N=5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — No pneumothorax related to study procedure, was due to the rupture of an abscess secondary to aspiration, causing a bronchopleural fistula
altered mental state (General disorders) | 0 | 2 — Not related to study; documented ICU delirium due to hospitalization for underlying disease, causing waxing and waning of consciousness.
unplanned readmission (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Unrelated to study; patient readmitted for syncope, found to have non-occlusive pulmonary thrombus after being discharged from index hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Operative VATS Decortication (N=5) | Non-operative Fibrinolytic Therapy (N=5)
additional CT (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — Subjects needed additional imaging

LIMITATIONS AND CAVEATS:
Potential limitations to this study include a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT03583931/Prot_SAP_000.pdf